CLINICAL TRIAL: NCT01458236
Title: A Multinational, Multicenter, Double-blind, Randomized, Placebo-controlled, Phase III Study to Assess the Efficacy and Safety of BPS-314d-MR in Subjects With Pulmonary Arterial Hypertension Currently Receiving Treatment With an Endothelin Receptor Antagonist and/or a Phosphodiesterase-5 Inhibitor
Brief Title: A Multinational, Multicenter, Study to Assess the Efficacy and Safety of BPS-314d-MR in Subjects With Pulmonary Arterial Hypertension Currently Receiving Treatment With an Endothelin Receptor Antagonist and/or a Phosphodiesterase-5 Inhibitor
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Lung Biotechnology PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BPS-314d-MR-PAH-301
Record Dates: First submitted 2011-09-29; First posted 2011-10-24 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — beraprost

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BPS-314d-MR (Experimental): Available as 15 μg and 60 μg tablets for oral, twice daily (BID) administration.
  Interventions: Drug: Beraprost Sodium 314d Modified Release Tablets
- Placebo (Experimental): Placebo tablets, which are identical in size and appearance to those containing BPS-314d-MR and are for oral, BID administration, will be utilized in subjects assigned to the placebo study drug treatment group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Beraprost Sodium 314d Modified Release Tablets — Available as 15 μg and 60 μg tablets for oral, twice daily (BID) administration
  Arms: BPS-314d-MR
Drug: Placebo — Placebo tablets, which are identical in size and appearance to those containing BPS-314d-MR and are for oral, BID administration, will be utilized in subjects assigned to the placebo study drug treatment group
  Arms: Placebo

SUMMARY:
A multinational, multicenter, double-blind, randomized, placebo-controlled, Phase III study to assess the efficacy and safety of BPS 314d-MR in subjects with pulmonary arterial hypertension currently receiving treatment with an Endothelin Receptor Antagonist (ERA) and/or a Phosphodiesterase-5 Inhibitor (PDE-5 inhibitor).

Approximately 100 centers will be participating in the study. Approximately 630 eligible subjects will be randomized 1:1 into two groups, BPS-314d-MR (active) or placebo study drug.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety of BPS-314d-MR in subjects with PAH who are treated with background therapy such as ERA and/or a PDE-5 inhibitor.

Subjects who consent to the study will be assessed at the Screening and Baseline visits to determine eligibility for the study. Subjects meeting eligibility criteria at the Baseline visit will be enrolled into the study and treated by either active or placebo study drug. The subject, the clinical site staff and the Sponsor will be blinded to the treatment assignment. Treatment assignment will be random.

Following the Baseline visit, subjects will return to the clinical site at Week 6, Week 12, Week 20 and every 12 weeks thereafter. Subjects will undergo all scheduled efficacy and safety assessments, as defined by the protocol. Between scheduled clinical site visits, the clinical site staff will be required to contact the subject by a telephone call to assess tolerability to study drug and change subject's dosage as appropriate. Telephone calls should occur at least once weekly for the first 20 study weeks when dose changes will occur most frequently and subjects are becoming familiar with the study procedures. Telephone calls will occur at least once monthly thereafter. Subjects will be provided with an electronic diary to record doses taken and help in tracking of health issues for conversations with the clinical site staff.

Subjects will continue their participation in the study until the Sponsor formally closes the study. At that time the subject will return to the clinical site for an End of Treatment visit to complete all scheduled tests. Subjects who are participating in the study at its conclusion may be offered the opportunity to enroll in a long-term extension study. Subjects who do not continue into an extension study are required to discontinue from study drug.

Subjects will be urged to remain in the study for long-term follow-up even if study drug is discontinued.

In the event that a subject withdraws consent for participation in the study or the Investigator terminates the subject from the study the subject will return to the clinical site for an End of Treatment visit to complete all scheduled tests. After study drug has been permanently discontinued, and if the subject is terminated from the study, the subject will return to the clinical site after 30-37 days for a final Safety Follow-up visit and to return any remaining study drug.

The optional Pharmacokinetic (PK) evaluation will be offered to all study subjects at clinical sites. Subjects within those sites will decide if they wish to participate in the optional PK evaluation. For those subjects electing to participate, two blood samples will be collected at three clinical site visits (Weeks 6, 12 and 20).

The optional hemodynamic sub-study will be offered to all study subjects at clinical sites. All subjects at the selected research centers will be offered the opportunity to volunteer in the sub-study. Hemodynamic measurements will be assessed by Right Heart Catheterization (RHC). For those subjects who consent to the RHC, the RHC procedure will be performed at the Baseline visit and during Week 20.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 80 years (inclusive).
2. Established diagnosis of pulmonary arterial hypertension that is either idiopathic or familial PAH, collagen vascular disease associated PAH, PAH induced by anorexigens/toxins, or PAH associated with repaired congenital systemic-to-pulmonary shunts (repaired ≥5 years).
3. Clinically stable PAH as determined by the Investigator.
4. Able to walk unassisted (oxygen use allowed).
5. A 6-Minute Walk distance (6MWD) of 150 to 450 meters (inclusive) at Screening.
6. A 6MWD at the Baseline visit that is within 15% of the Screening 6MWD.
7. An average 6MWD (Screening and Baseline visits) of 150 to 450 meters (inclusive).
8. Previous (within five years prior to the Baseline visit) right heart cardiac catheterization (RHC) with findings consistent with PAH, specifically mean Pulmonary Arterial Pressure (PAPm) ≥25 mmHg (at rest), Pulmonary Capillary Wedge Pressure (PCWP) (or left ventricular end diastolic pressure) ≤15 mmHg, and Pulmonary Vascular Resistance (PVR) >3 mmHg/L/min.
9. Previous (within five years prior to the Baseline visit) chest radiograph consistent with the diagnosis of PAH.
10. Has been on a current background regimen of an ERA and/or PDE-5 inhibitor for a minimum of 90 days with at least 30 days on a stable dose of ERA and/or PDE-5 inhibitor prior to the Baseline visit.
11. Women of child-bearing potential (defined as less than 1 year post-menopausal and not surgically sterile) must be practicing abstinence or using two highly effective methods of contraception (defined as a method of birth control that result in a low failure rate, i.e., less than 1% per year, such as approved hormonal contraceptives, barrier methods [such as a condom or diaphragm] used with a spermicide, or an intrauterine device). Subject must have a negative pregnancy test at the Screening and Baseline visits.
12. Willing and able to comply with study requirements and restrictions.

Exclusion Criteria:

1. Has pulmonary venous hypertension, pulmonary veno-occlusive disease, pulmonary capillary hemangiomatosis, or chronic thromboembolic pulmonary hypertension.
2. As the diagnosis of PAH may be challenging in subjects with multiple co-morbid conditions, if the subject has the presence of two or more of the following co-morbid conditions:

   * Diabetes
   * Age > 70 years
   * Body Mass Index [BMI] > 35
   * Past history of pulmonary embolism
   * Chronic atrial fibrillation
   * FEV1 of < 70% of predicted
   * Systemic hypertension requiring treatment. AND
   * the Sponsor does not concur, in writing, with the appropriateness of the subject to enter the study.
3. Has a history of interstitial lung disease, unless subject has collagen vascular disease and has had pulmonary function testing conducted within 6 months of the Baseline visit demonstrating a total lung capacity ≥70% of predicted.
4. Has a history of obstructive lung disease, unless subject has had pulmonary function testing conducted within 6 months of the Baseline visit demonstrating a forced expiratory volume in 1 second (FEV1) of ≥ 50% of predicted.
5. Is pregnant or lactating.
6. Has received prostanoid therapy at any time.
7. Modified dose, initiated or discontinued any PAH medication within 30 days prior to the Baseline visit including, but not limited to, an ERA, PDE-5 inhibitor, oral vasodilators, diuretics, digoxin, oxygen or calcium channel blocker (with the exception of anticoagulants).
8. Has an ongoing hemorrhagic condition (e.g., upper digestive tract hemorrhage, hemoptysis, etc.), or has a pre existing condition that, in the Investigator's judgment, may increase the risk for developing hemorrhage during the study (e.g., hemophilia). Transient hemorrhage (e.g., epistaxis, normal menstrual bleeding, gingival bleeding, hemorrhoidal bleeding, etc.) will not preclude enrollment
9. Has received any investigational medication, device or therapy within 30 days prior to the Baseline visit or is scheduled to receive another investigational drug, device or therapy during the course of the study.
10. Has any preexisting disease known to cause pulmonary hypertension other than those listed in the Inclusion Criteria.
11. Has any musculoskeletal disease or any other disease that would significantly limit ambulation.
12. Has any form of unrepaired or recently repaired (< 5 years) congenital systemic-to-pulmonary shunt other than patent foramen ovale.
13. Documented history or current evidence of ischemic heart disease.
14. History of left sided myocardial disease as evidenced by a mean PCWP (or a left ventricular end diastolic pressure) > 15 mmHg or left ventricular ejection fraction < 40% as assessed by either multigated angiogram, angiography or echocardiography, or left ventricular shortening fraction <22% as assessed by echocardiography. Note that subjects in whom abnormal left ventricular function is attributed entirely to impaired left ventricular filling due to the effects of right ventricular overload (i.e., right ventricular hypertrophy and/or dilatation) will not be excluded.
15. Has creatinine clearance <30 (using the Crockroft-Gault formula) or requires hemodialysis.
16. Has Childs-Pugh class C liver cirrhosis.
17. Has had previous atrial septostomy.
18. Any other clinically significant illness that, in the opinion of the Investigator, might put the subject at risk of harm during the study or might adversely affect the interpretation of the study data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Time-to-clinical-worsening | up to 252 weeks
  Clinical worsening events:
  * All-cause death
  * Non-planned PAH-related hospitalization (i.e. for at least 24 hours caused by a clinical condition related to PAH such as right heart failure, arrhythmia, syncope, hemoptysis, chest pain or dyspnea).
  * Addition of parenteral (i.e. IV or SQ) prostanoid therapy
  * ≥15% decrease from baseline in 6MWD, confirmed by 2 consecutive tests performed 1 to 28 days apart
  * Increase from Baseline Visit in WHO functional class

SECONDARY OUTCOMES:
World Health Organization Functional Class (WHO) | up to 252 weeks
  The outcome will be measured at baseline (Day 1) and at each visit (From baseline to week 6 visit, to week 12 visit, to week 20 visit, to quaterly follow up visits, to End of treatment visit)
Borg Dyspnea Score | up to 252 weeks
  The outcome will be measured at baseline (Day 1) and at each visit (From baseline to week 6 visit, to week 12 visit, to week 20 visit, to quaterly follow up visits, to End of treatment visit)
pro-BNP levels (Pro-B Type Brain Natriuretic Peptide) | up to 252 weeks
  The outcome will be measured at baseline (Day 1) and at each visit (From baseline to week 6 visit, to week 12 visit, to week 20 visit, to quaterly follow up visits, to End of treatment visit)
6 Minute Walk Distance (6MWD) | up to 252 weeks
  The outcome will be measured at baseline (Day 1) and at each visit (From baseline to week 6 visit, to week 12 visit, to week 20 visit, to quaterly follow up visits, to End of treatment visit)